CLINICAL TRIAL: NCT04634227
Title: A Pilot Study of Gemcitabine Plus High-Dose Ascorbate in Locally Advanced Unresectable or Metastatic Soft Tissue and Bone Sarcomas in Adults
Brief Title: Gemcitabine Plus Ascorbate for Sarcoma in Adults (Pilot)
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Mohammed Milhem, MBBS (Other)
Responsible Party: Principal Investigator, John Rieth, Clinical Assistant Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201802800 (Pilot)
Record Dates: First submitted 2020-11-16; First posted 2020-11-18 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Sarcoma; Soft Tissue Sarcoma; Unresectable Soft Tissue Sarcoma; Metastatic Bone Tumor; Bone Sarcoma
Keywords: Sarcoma; Soft tissue; Ascorbate
MeSH Terms: conditions — Sarcoma; Bone Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemcitabine + High-Dose Ascorbate (Experimental): Ascorabte is administered on Days 1, 2, 8, 9, 15 and 16 of a 28-day cycle. Gemcitabine will be administered on Days 1, 8 and 15, after the infusion of ascorbate. Concomitant treatment will continue for 6 cycles. Patients whose disease has not progressed while receiving gemcitabine and ascorbate and who are tolerating therapy may continue either single agent gemcitabine or concomitant treatment beyond 6 cycles at the discretion of the investigator. Treatment will be terminated with progression of disease. Disease will be assessed by CT of the chest, abdomen and pelvis or MRI of the lesion every 2 cycles for progression.
  Interventions: Drug: Ascorbate

INTERVENTIONS:
Drug: Ascorbate — Following 15g test dose, 75g administered 75g dose on days 1 and 2. Further doses of ascorbate will be determined by serum ascorbate levels measured by the end of the week to reach a target serum concentration between 20 -30 mM. Ascorbate doses will continue to be escalated until either the target serum concentration or maximum dose of 125 g is administered.

SUMMARY:
This study will enroll patients who have a diagnosis of locally advanced, unresectable or metastatic soft tissue or bone sarcoma (except gastrointestinal stromal tumors and Kaposi's sarcoma) from any site.

DETAILED DESCRIPTION:
The primary objectives of this pilot study are to assess the feasibility of pharmacokinetically-guided, patient-individualized dosing and to obtain preliminary evidence of anti-tumor activity of intravenous ascorbate in combination with gemcitabine to inform a subsequent Phase II trial. Soft tissue and bone sarcomas will be studied as different cohorts given the differences in biology and historical responses to single agent gemcitabine in these disease types. As such, 10 evaluable patients per disease cohort will be included.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years old
* ECOG Performance Status of ≤ 2
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Tolerate a 15g ascorbate infusion (screening dose)
* Any patient with the diagnosis of locally advanced, unresectable or metastatic soft tissue or bone sarcoma (except GIST and Kaposi's) from any site. A minimum of 1 prior chemotherapy regimen, including adjuvant or neo-adjuvant therapy for the treatment of sarcoma. Patients eligible for an anthracycline should have received a prior anthracycline containing regimen. Patients who decline or are not eligible for anthracycline treatment may be considered for this protocol as a first line treatment. Patients with a diagnosis of liposarcoma should also have received eribulin if they received anthracycline-based therapy prior to eribulin. Patients with a diagnosis of myxoid liposarcoma should have received trabectedin. Patients with angiosarcoma should have received either taxol or docetaxel. Patients must have measurable disease defined as at least 1 lesion ≥ 1cm in the greatest dimension.
* Patients with metastatic bone sarcomas who have failed all available therapies that have demonstrated clinical benefit. Available therapies include but not limited to methotrexate, adriamycin and cisplatin for osteosarcoma and vincristine, adriamycin and Cytoxan, ifosfamide, etoposide (VAC/IE) for Ewing's sarcoma.
* Patients must have had disease progression on or following their most recent treatment regimen or on presentation for the first time with locally advanced unresectable or metastatic disease.
* Patients with NO known CNS disease, except for treated brain metastasis: Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded

Exclusion Criteria:

* Lab values in the below ranges:

  * Neutrophil count of </=1500/mm3
  * Platelet count of </= 100,000/mm3L
  * Hemoglobin < 9 g/dL (transfusion to meet eligibility allowed)
  * AST/SGOT and ALT/SGPT > 2.5 x upper limit of normal (ULN) or >5.0 x ULN if the transaminase elevation is due to disease involvement
  * Alkaline phosphatase > 5 x ULN without known bony metastases
  * Serum bilirubin >1.5 x ULN
  * Serum creatinine > 1.5 x ULN or 24-hour creatinine clearance <50 ml/min
  * Total serum calcium < LLN or if calcium is below LLN then corrected calcium for serum albumin should be >/= LLN
  * Serum potassium < 3.0
  * Serum sodium < 130
  * Serum albumin <2.5g/dl
* G6PD (glucose-6-phosphate dehydrogenase) deficiency
* Prior exposure to gemcitabine for metastatic disease
* Subjects with prior doxorubicin exposure with a MUGA or ECHO demonstrating LVEF < the lower limit of the institutional normal.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Actively receiving insulin or requiring fingerstick glucose monitoring at time of ascorbate infusion
* Patients on warfarin and unable to be substituted to another anticoagulant
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Pregnancy (positive pregnancy test) or lactation.
* Women of childbearing potential (WOCBP) who are not willing to use two methods of contraception one of them being a barrier method during the study and for 3 months after last study drug administration
* Patients who are on the following drugs and cannot have a drug substitution: flecainide, methadone, amphetamines, quinidine, and chlorpropamide. High dose ascorbic acid may affect urine acidification and, as a result, may affect clearance rates of these drugs.
* Other concurrent severe and/or uncontrolled medical conditions
* Patients who have received chemotherapy or any investigational drug < 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study.
* Concomitant use of any other anti-cancer therapy or radiation therapy. Palliative radiation therapy to non-target lesions is permitted.
* Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom.
* Patients with a history of another primary malignancy within 2 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin
* Patients with known positivity for human immunodeficiency virus (HIV); baseline testing for HIV is not required. High-dose ascorbate acid is a known CYP450 3A4 inducer, which results in lower serum levels of antiretroviral drugs.37
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
* Patients with history of more than one symptomatic oxalate stone in the last 6 months or visible stone in the kidney or ureter on screening CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the 12 weeks progression free survival (PFS 12) at 12 weeks post treatment initiation | 12 weeks post-treatment
  The primary endpoint of interest is PFS12 defined as the proportion of patients without progressive disease per RECIST 1.1 at 12 weeks after treatment initiation. A sample size of 10 evaluable patients per disease cohort (soft tissue and bone) will allow for the estimation of PFS12 per the 90% exact confidence intervals as follows:
  PFS12 Exact 90% confidence interval:
  1/10 10% (1-39%); 2/10 20% (4-51%); 3/10 30% (9-61%); 4/10 40% (15-70%); 5/10 50% (22-78%); 6/10 60% (30-85%); 7/10 70% (39-91%); 8/10 80% (49-96%); 9/10 90% (61-99%);

SECONDARY OUTCOMES:
Assess overall survival of patients with unresectable or metastatic soft tissue and bone sarcoma treated with high dose ascorbate when administered intravenously concurrently with gemcitabine | Every 2 months for first 6 months, then every 3 months up to 2 years post treatment
  Time from start of therapy (day 1, cycle 1) to death.
Determine the tumor response as per RECIST 1.1 criteria | 12 weeks post-treatment
  Tumor response will be defined using the RECIST 1.1 guidelines as below
  * Complete response is the disappearance of all target lesions; Any pathological lymph nodes ( whether target or Non-target) must have reduction in short axis to <10mm.
  * Partial response is a 30% decrease in the sum of the longest dimension (LD) of target lesions, relative to baseline measurement;
  * Progressive disease is an increase of 20% or more in the sum of the LD of target lesions, taking as reference the smallest sum on study. The sum must also demonstrate an absolute increase of at least 5 mm.Or appearance of a new malignant lesion.
  * Stable disease is a decrease in tumor size of less than 30% or increase of less than 20%.
Incidence of Adverse Events (AE) Per CTCAE 4.03 | Up to 30 days after completion of study treatment
  Evaluate the safety and tolerability of this regimen by the incidence of AEs per CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: John Rieth, MD, Principal Investigator — University of Iowa Hospitals & Clinics
Locations (1):
- John, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No